CLINICAL TRIAL: NCT00205569
Title: Acute Cognitive and Neurobehavioral Intervention: Efficacy Evaluation (a Research Project Within the Traumatic Brain Injury Model System Grant)
Brief Title: Acute Cognitive and Neurobehavioral Intervention: Efficacy Evaluation
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H133A02051603; H133A020516
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Traumatic Brain Injury
Keywords: brain injury, acute rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Individuals with traumatic brain injury requiring inpatient rehabilitation.
  Interventions: Behavioral: First Steps Educational Curriculum

INTERVENTIONS:
Behavioral: First Steps Educational Curriculum — 10 sessions with the research participant to review an educational curriculum regarding brain injury rehabilitation and community reintegration

SUMMARY:
To learn more about behavior and everyday functioning after brain injury, and to learn if behavior and functioning gets better with more education about changes after brain injury.

DETAILED DESCRIPTION:
To evaluate the efficacy of the First Steps intervention for improving neurobehavioral functioning, functional status, and life satisfaction, and for increasing knowledge about TBI and compensatory strategies. The First Steps program was developed to address the neurobehavioral and emotional concerns of survivors of TBI during the course of inpatient rehabilitation. Program format and content reflects clinical experience and extensive research review. Input from survivors, family members, and rehabilitation staff trained in working with the TBI population has also helped shape the implementation protocol. The foundation of the protocol is a curriculum [Niemeier, J., Kreutzer, J., & Taylor, L. (2005). Acute cognitive and neurobehavioral intervention for individuals with acquired brain injury: Preliminary outcome data. Neuropsychological Rehabilitation, 15(2), 129-146.] The First Steps curriculum consists of ten lessons and was developed to address the common needs, issues, and concerns of TBI survivors admitted acutely for inpatient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* adults (18 years or older) who have experienced a TBI (damage to brain tissue caused by an external mechanical force as evidenced by: loss of consciousness due to brain trauma, or post traumatic amnesia, or skull fracture, or objective neurological findings that can be reasonably attributed to TBI on physical examination or mental status examination).

Exclusion Criteria:

* imminent risk of psychiatric hospitalization, or in imminent danger of hurting themselves or others.
* unable to tolerate treatment sessions due to physical, cognitive, behavioral, or other difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with traumatic brain injury requiring inpatient rehabilitation and admitted to Virginia Commonwealth University's Medical College of Virginia Hospitals acutely after injury.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2002-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Kreutzer, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Result] Niemeier JP, Kreutzer JS, Taylor LA. Acute cognitive and neurobehavioural intervention for individuals with acquired brain injury: preliminary outcome data. Neuropsychol Rehabil. 2005 May;15(2):129-46. doi: 10.1080/09602010443000083. PMID 16353506